CLINICAL TRIAL: NCT06499818
Title: Circumferential Pulmonary Vein Isolation Alone Versus CPVI Plus Low-Voltage Areas Ablation During SR Versus CPVI Plus Low-Voltage Areas Ablation During AF for the Treatment of CAF
Brief Title: CPVI Alone Versus CPVI Plus Low-Voltage Areas Ablation During SR Versus CPVI Plus Low-Voltage Areas Ablation During AF for the Treatment of CAF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yantai Yuhuangding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-226
Record Dates: First submitted 2024-07-07; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STABLE-SR (Experimental)
  Interventions: Procedure: STABLE-SR
- STABLE-AF (Experimental)
  Interventions: Procedure: STABLE-AF
- CPVI alone (Active Comparator)
  Interventions: Procedure: CPVI

INTERVENTIONS:
Procedure: STABLE-SR — homogenization of the low voltage zones and elimination of the complex electrograms from the transitional zones during sinus rhythm
  Arms: STABLE-SR
Procedure: STABLE-AF — homogenization of the low voltage zones and elimination of the complex electrograms from the transitional zones during Atrial Fibrillation
  Arms: STABLE-AF
Procedure: CPVI — ablate around the pulmonary vein orifice
  Arms: CPVI alone

SUMMARY:
The primary objective of this investigation is to compare the efficacy of Three different AF ablation strategies in patients with Persistent atrial fibrillation: CPVI plus Low-Voltage Areas ablation during sinus rhythm Versus. CPVI Plus Low-Voltage Areas Ablation During AF and CPVI alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age is 18-80 years;
2. Patients with non-paroxysmal AF; non-paroxysmal AF will be defined as a sustained episode lasting > 7 days;
3. Patients can sign the written informed consent for the study;
4. Patients can endure the required follow-up.

Exclusion Criteria:

1. Patients who had previously undergone atrial fibrillation, atrial tachycardia, or atypical atrial flutter ablation
2. Preoperative combined atrial tachycardia (≥30S) and atypical atrial flutter
3. Left atrial diameter >55mm
4. Left ventricular ejection fraction <35%
5. Left atrial thrombus
6. Postoperative cardiac surgery
7. After valve replacement
8. After permanent pacemaker implantation
9. hypertrophic cardiomyopathy
10. Patients with moderate-to-severe aortic valve disease, moderate-to-severe mitral stenosis, and severe other valvular disease
11. Hemorrhagic stroke within 6 months
12. Transient ischemic attack or ischemic stroke within 1 month
13. Mental disorder or history of mental illness and inability to cooperate voluntarily
14. Breastfeeding, pregnancy and women planning or likely to become pregnant
15. Life expectancy <12 months
16. Participating in other interventional clinical trials
17. The researchers judged that it was not suitable for inclusion in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of no atrial arrhythmias greater than 30 seconds | at least 18 months follow up
  The incidence of no atrial arrhythmias greater than 30 seconds

SECONDARY OUTCOMES:
No use of antiarrhythmic drugs and no occurrence of atrial fibrillation exceeding 30 seconds | at least 18 months follow up
  No use of antiarrhythmic drugs and no occurrence of atrial fibrillation exceeding 30 seconds
No use of antiarrhythmic drugs and no occurrence of atrial tachycardia/flutter exceeding 30 seconds | at least 18 months follow up
  No use of antiarrhythmic drugs and no occurrence of atrial tachycardia/flutter exceeding 30 seconds
Atrial fibrillation load | at least 18 months follow up
  Atrial fibrillation load
Procedure time | Surgical procedure
  time that the patient spend in the procedure room
Ablation time | 1 week after patient enrollment
  the total Ablation time, during CPVI and after CPVI
Incidence of peri-procedural complications | at least 18 months follow up
  stroke, PV stenosis, cardiac perforation, esophageal injury and death

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT06499818/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT06499818/ICF_001.pdf